CLINICAL TRIAL: NCT01937052
Title: Johns Hopkins Breast Cancer Program Hormone Therapy Longitudinal Database
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: J1189; SKCCC J1189 (Other: SKCCC at Johns Hopkins); NA_00051923 (Other: JHM IRB)
Record Dates: First submitted 2013-09-03; First posted 2013-09-09 (Estimated); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Specimen Handling; Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (for example: serum, plasma, and whole blood) and saliva samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast cancer patients: All patients planned to initiate hormonal therapy with either Tamoxifen, Raloxifene (Evista®), Anastrozole (Arimidex®), Letrozole (Femara®) or Exemestane (Aromasin®) are eligible to participate in sample collection and data for patient-reported outcomes/questionnaires.
  Interventions: Other: Sample collection; Behavioral: Patient-reported outcomes

INTERVENTIONS:
Other: Sample collection — Participants will be offered the option to consent for blood (preferred) or saliva for DNA pharmacogenetic testing, and for additional samples for banking for future studies.
Behavioral: Patient-reported outcomes — Patient reported outcomes (PROs) will be collected via electronic questionnaires that will be administered to patients at regular intervals per the study calendar; in most cases, this should coincide with medical oncology follow-up.

SUMMARY:
The purpose of this project is to establish a repository of information and samples from breast cancer patients or those at high risk of developing breast cancer, who are initiating hormone therapy as part of standard clinical care or prevention. This repository will include patient reported outcomes and other questionnaires, information on medication use, data about adherence to the hormone therapy and tumor characteristics, including prospectively collected samples.

DETAILED DESCRIPTION:
This research is being done to learn more about the side effects of breast cancer hormone therapy and if a person's genetic information may help us to develop a way to predict the side effects a patient may have and how best to treat them. In addition, the investigators hope to look at how the side effects from hormone therapy influence a patient's willingness to continue hormonal treatment.

Men and women being prescribed hormone therapies including Tamoxifen, Raloxifene (Evista), Anastrozole (Arimidex), Letrozole (Femara), or Exemestane (Aromasin), by their oncologist for either prevention of breast cancer or treatment of breast cancer may join.

The decision of which hormone therapy to receive is the decision of the patient and physician, this study will collect samples and patient-reported outcomes during this routine, standard of care and will not direct any treatment decisions or interventions in any way.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 years of age or older
* Physically and cognitively able to complete the questionnaires
* Meet one of the following categories: 1) Initiating hormonal therapy for breast cancer prevention. All patients planned to initiate hormonal therapy with either Tamoxifen, Raloxifene (Evista®), Anastrozole (Arimidex®), Letrozole (Femara®) or Exemestane (Aromasin®) are eligible; concomitant use of Zoladex or Lupron is permitted; 2) Patients with histologically proven ductal carcinoma in situ (DCIS/stage 0) or stage I-III invasive carcinoma of the breast that is estrogen (ER) and/or progesterone (PR) positive by immunohistochemical staining, who are considering one of the above listed SERMs or AIs. These patients must have completed any planned chemotherapy and local therapy (e.g., lumpectomy or mastectomy); however, enrollment/initiation of hormonal therapy on study may be done prior to completion of radiation and/or biologic therapy (e.g., trastuzumab) at the discretion of the treating team; or, 3) The patient is aware of the nature of her diagnosis, understands the study regimen, its requirements, risks, and discomforts, and is able and willing to sign an informed consent form.
* Patients transitioning from one hormonal agent listed above to another may be enrolled prior to initiation of the new medication.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women being prescribed hormone therapies including Tamoxifen, Raloxifene (Evista), Anastrozole (Arimidex), Letrozole (Femara), or Exemestane (Aromasin), by their oncologist for either prevention of breast cancer or treatment of breast cancer may join.
Sampling Method: Non-Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2012-05-09 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Sample and data collection | 10 years
  To collect high quality prospective data regarding individual genetic profiles, medication use and patient reported outcomes on hormone therapy, which can be used to validate correlations that have been observed in other studies.

CONTACTS AND LOCATIONS:
Overall Officials: Vered Stearns, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Uhelski AR, Blackford AL, Sheng JY, Snyder C, Lehman J, Visvanathan K, Lim D, Stearns V, Smith KL. Factors associated with weight gain in pre- and post-menopausal women receiving adjuvant endocrine therapy for breast cancer. J Cancer Surviv. 2024 Oct;18(5):1683-1696. doi: 10.1007/s11764-023-01408-y. Epub 2023 Jun 1. PMID 37261654
- [Derived] Verma N, Blackford AL, Thorner E, Lehman J, Snyder C, Stearns V, Smith KL. Factors associated with worsening sexual function during adjuvant endocrine therapy in a prospective clinic-based cohort of women with early-stage breast cancer. Breast Cancer Res Treat. 2022 Dec;196(3):535-547. doi: 10.1007/s10549-022-06750-w. Epub 2022 Oct 5. PMID 36197536